CLINICAL TRIAL: NCT06450925
Title: A Randomized Double Blinded Trial of Vitamin A Supplementation in Allogeneic Stem Cell Transplantation.
Brief Title: Vitamin A Supplementation in Allogeneic Stem Cell Transplantation.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-0301
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Graft Vs Host Disease; Vitamin A Deficiency; Vitamin D Deficiency
MeSH Terms: conditions — Graft vs Host Disease; Vitamin A Deficiency; Vitamin D Deficiency | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin A (Active Comparator): Route of administration: Oral. Frequency: Once. Timing: Pre-transplant Dose of Vit A: 1.2 mg/kg, max dose 75 mg Formulation of Vit A: 2.5 mg liquid filled oral capsules.
  Vitamin A level assessment: Vitamin A levels will be measured pre-transplant and again at day +30 (± 10 days)
  Interventions: Drug: Vitamin A
- Placebo (Placebo Comparator): Placebo pills containing microcrystalline cellulose will be dispensed in patients who are randomized to the placebo arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin A — Enrolled subjects will receive one observed oral vitamin A dose, prior to their HSCT, in the outpatient clinic or inpatient Bone Marrow Transplant (BMT) floor.
  Arms: Vitamin A
Other: Placebo — Placebo pills containing microcrystalline cellulose will be dispensed in patients who are randomized to the placebo arm.
  Arms: Placebo

SUMMARY:
The investigators hypothesize that single oral high dose supplementation with vitamin A will reduce the incidence of moderate-severe chronic graft-versus-host disease (GVHD) compared with placebo.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is an effective treatment strategy for many malignancies, marrow failure syndromes, and immune deficiencies in children, adolescents, and adults. Vitamin A and its derivatives regulate growth and differentiation of intestinal cells, and vitamin A deficiency is associated with increased susceptibility to infection in both human and animal models. The investigators' preliminary data suggest lower vitamin A levels were associated with an increased incidence of gastrointestinal graft versus host disease (GI GVHD) in patients undergoing HSCT.

This study is a randomized double blinded comparison of vitamin A supplementation comparing a single large dose of vitamin A with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Be scheduled for allogeneic stem cell transplant.
* Have a vitamin A level < upper limit of normal for age.
* Be able to tolerate enteral vitamin dose administration.
* Have a total bilirubin level < 1.5x ULN and an AST and/or ALT< 3xULN for age
* Receiving PBSCs as stem cell graft

Exclusion Criteria:

* Ongoing raised intracranial pressure
* Liver cirrhosis
* Patients will be excluded if they are currently pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate-severe chronic graft versus host disease (GVHD) | 1 year after transplant
  Incidence of moderate-severe chronic GVHD

SECONDARY OUTCOMES:
Incidence of acute gastrointestinal graft versus host disease (GI GVHD) | 2 years after transplant
  Incidence of acute GI GVHD
Incidence of relapse | 2 years after transplant
  Incidence of relapse
Overall survival. | 2 years after transplant
  Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Khandelwal, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - The Ohio State University, Columbus, Ohio